CLINICAL TRIAL: NCT05153616
Title: Periodic Limb Movements Among Dialysis and Non-dialysis Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Samah Kotb Mohamed, Aswan University Hospital, Aswan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 150/7/17
Record Dates: First submitted 2021-11-28; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: The Aim of the Study Was to Screen Prevalence of Periodic Limb Movements Among Chronic Kidney Disease Patients
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Polysomnography (Experimental)
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Full night attended polysomnography to diagnose periodic limb movements

SUMMARY:
Periodic leg movement disorder is defined as periodic episodes of repetitive limb movements during sleep that mainly occur in the lower limb, including the hips, knees and toes and sometimes affects the upper limb. It may be accompanied by frequent nocturnal arousals, and if so, this sleep disturbance may cause excessive daytime sleepiness. Chronic kidney disease patients are at risk of periodic leg movements and common causes are iron deficiency, anemia, raised serum calcium and central and peripheral nervous system disorders.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease

Exclusion Criteria:

* diabetic, hepatic and chrest disease patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Periodic limb movement | One night
  Screening the prevalence of periodic limb movement

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No